CLINICAL TRIAL: NCT01943201
Title: Does a Low Friction Bed Sheet Optimize the Skin, Resistance and Physiology and Reduce the Risk for Pressure Ulcer?
Brief Title: Low Friction Bed Sheet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Collaborators: Swiss Federal Laboratories for Material Sciences and Technology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2010-04
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Spinal Cord Injury; Pressure Ulcer
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- new bedsheet (Experimental): new bedsheet
  Interventions: Device: new bedsheet
- conventional bedsheet (Placebo Comparator): conventional bedsheet
  Interventions: Device: conventional bedsheet

INTERVENTIONS:
Device: new bedsheet — sleeping 5 nights on the new bedsheet
  Other Names: specially developed low-friction hospital bed sheet
  Arms: new bedsheet
Device: conventional bedsheet — sleeping 5 nights on the conventional bedsheet
  Other Names: normal hospital bedsheet
  Arms: conventional bedsheet

SUMMARY:
Introduction:

It is known that people with spinal cord injury (SCI) bear a considerably increased risk of developing pressure ulcer, whereby frictional forces and shear forces are recognized as risk factors. It was the aim of the study to examine the effects of a specially developed low-friction hospital bed sheet on skin physiology as well as it's acceptance by patients with SCI.

Method:

Prospective, randomised crossover study. Patients with a subacute spinal cord injury will be recruited. Each patient spends five consecutive nights on the new, respectively, conventional bed sheet. After the five nights, patients are asked to complete a linear questionnaire (VAS) concerning well-being, odour, perspiration and wrinkling. In addition, the patients are examined daily while still fasting, for skin redness, skin moisture, skin elasticity and skin blood circulation in the parasacral region.

ELIGIBILITY:
Inclusion Criteria:

* SCI patients without a presser ulcer for the last 2 months
* Paraplegic and tetraplegic patients
* complete and incomplete lesion (AIS A, AIS B, AIS C, AIS D)
* caused by illness or traumatic event
* smoker and non-smoker

Exclusion Criteria:

* progressive disease
* severe accessory symptoms (diabetes mellitus, coronary heart disease, severe renal failure)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
well-being | 1 day in the morning after sleeping on the new bed sheet
  linear questionnaire (visual analogue scale)

SECONDARY OUTCOMES:
Skin redness | 1 day in the morning after sleeping on the new bed sheet
  Measurement: Mexameter 10 points of measurement in the sacral region
Skin perfusion | 1 day in the morning after sleeping on the new bed sheet
  Measurement: PeriFlux 10 points of measurement in the sacral region
Skin hydration | 1 day in the morning after sleeping on the new bed sheet
  Measurement: Corneometer 10 points of measurement in the sacral region
Skin elasticity | 1 day in the morning after sleeping on the new bed sheet
  Measurement: Cutometer 10 points of measurement in the sacral region

CONTACTS AND LOCATIONS:
Overall Officials: Anke Scheel, MD, Principal Investigator — Swiss Paraplegic Center
Locations (1):
- Swiss Paraplegic-Centre, Nottwil, Canton of Lucerne, Switzerland

REFERENCES:
- See also: Swiss Paraplegic Centre Nottwil — http://www.paraplegie.ch